CLINICAL TRIAL: NCT04109833
Title: Impact of Early Antibiotic Therapy on Vaccination Response in Preterm Infants
Brief Title: Early Antibiotic Therapy and Vaccination
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Natascha Köstlin-Gille, Junior Research Group Leader, University Hospital Tuebingen
Other Study IDs: 368/2019BO1
Record Dates: First submitted 2019-09-27; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Vaccination Reaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — stool samples for microbiome analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- no antibiotic therapy (ABT) in the first week of life: VLBWI with gestational age between 24+0 and 28+6 weeks of gestation without antibiotic treatment in the first week of life
- ABT in the first week of life: VLBWI with gestational age between 24+0 and 28+6 weeks of gestation with antibiotic treatment in the first week of life
  Interventions: Drug: ABT

INTERVENTIONS:
Drug: ABT — any antibiotic therapy in the first week of life
  Other Names: any antibiotic therapy
  Groups: ABT in the first week of life

SUMMARY:
Neonatal Sepsis is one of the most common causes of death in preterm infants. Therefore, up to 80% of very low birth weight infants receive antibiotic therapy in their first week of life. Antibiotic therapy is one of the most important influencing factors for the establishment of the intestinal microbiome, which in turn modulates neonatal immune development. In this pilot study, it will be investigated, if antibiotic therapy in the first week of life influences the vaccination response of preterm infants.

DETAILED DESCRIPTION:
The aim of the study is to compare antibody titers against Hepatitis B, Polio, Pertussis, Haemophilus influenza B, Tetanus, Diphteria and Pneumococcus in very low birth weight infants (VLBWI) infants who received antibiotic therapy in their first week of life and who did not. In this pilot study, 20 VLBWI infants will be included (10 per group). Infants will be matched fo age and gender.

ELIGIBILITY:
Inclusion Criteria:

* born at University Hospital Tübingen
* at least one dose of antibiotics within the first week of life

Exclusion Criteria:

* genetic disorders
* chronic infections
* hematological disorders
* immunoglobulins within the first 60 days of life
* immunological disorders
* infants from Hepatitis B positive mothers

Ages: 24 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: preterm infants with gestational age between 24+0 and 28+6 weeks of gestation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-09-27 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
vaccination reaction | 7 months
  measurement of antibody titers for Hepatitis B, Polio, Pertussis, Haemophilus Influenza B, Tetanus, Diphteria and Pneumococcus 4 months after the first vaccination (at an age of 6 months)

SECONDARY OUTCOMES:
Microbiome composition | 7 months
  microbiome analyses of stool samples at age 14 days and corrected 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Natascha Köstlin-Gille, Dr. med., Principal Investigator — Department for Neonatology at University Hospital Tübingen
Locations (1):
- University Hospital, Tübingen, Baden-Wurttemberg, Germany